CLINICAL TRIAL: NCT02195453
Title: A Randomized,Double-blind,Placebo-Controlled,Multicenter Clinical Trail of Chemotherapy Combined With Yangzhengxiaoji Capsule in Patients With Advanced Non-Small Cell Lung Cancer
Brief Title: Chemotherapy Combined With Yangzhengxiaoji Capsule in Patients With Advanced Non-Small Cell Lung Cancer
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shandong Cancer Hospital and Institute (Other)
Collaborators: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Jinming Yu, Shandong Cancer Hospital and Institute, Shandong Cancer Hospital and Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: yl-yxb08-lcsyfa-201302
Record Dates: First submitted 2014-07-07; First posted 2014-07-21 (Estimated); Last update posted 2014-07-21 (Estimated); Status verified 2014-07

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Non-small cell lung cancer; FACT-L scale; Yangzhengxiaoji
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Yangzhengxiaoji Capsule (Experimental): Gemcitabine or Pemetrexed
  Cisplatin
  Yangzhengxiaoji Capsule four granules t.i.d po
  Interventions: Drug: Yangzhengxiaoji Capsule
- Placebo Capsule (Placebo Comparator): Gemcitabine or Pemetrexed
  Cisplatin
  Placebo Capsule four granules t.i.d po
  Interventions: Drug: Placebo Capsule

INTERVENTIONS:
Drug: Yangzhengxiaoji Capsule — Gemcitabine 1000mg/m² or Pemetrexed 500mg/m² IV drip on D1 and D8,21 days for a cycle.
  Cisplatin 75mg/m² IV drip for one day or two-three days total injection,21 days for a cycle.
  Yangzhengxiaoji Capsule four granules t.i.d po.
  Arms: Yangzhengxiaoji Capsule
Drug: Placebo Capsule — Gemcitabine 1000mg/m² or Pemetrexed 500mg/m²IV drip on D1 and D8,21 days for a cycle.
  Cisplatin 75mg/m² IV drip for one day or two-three days total injection, 21 days for a cycle.
  Placebo Capsule four granules t.i.d po.
  Arms: Placebo Capsule

SUMMARY:
The purpose of this study is to observe quality of life and treatment side effects in patients with advanced non small cell lung cancer (NSCLC) receive chemotherapy and Yangzhengxiaoji capsule.

ELIGIBILITY:
Inclusion criteria:

1. Histology and/or cytology confirmed stage Ⅳ NSCLC patients;
2. With at least one measurable solid tumor (RECIST standard version 1.1): tumor >=10 mm in diameter on CT or MRI images, or lymph node >=15 mm in diameter on CT or MRI images;
3. Eastern Cooperative Oncology Group(ECOG) score 0-1, expectant survival > 3 months;
4. Age: 18-70 years;
5. Normal organ function:

   Bone marrow: neutrophils (ANC) count>=1.5×10^9/L, Platelets count>=100×10^9/L, hemoglobin>=90g/L；Renal function, serum creatinine<=1.5 mg/dl, and/or creatinine clearance or>=60 ml/min; Liver function: total serum bilirubin levels <= 1.5 times the upper limit of normal (ULN), serum aspartate aminotransferase (AST) or serum alanine aminotransferase (ALT)<=2.5 times the ULN, if abnormal liver function caused by the underlying malignancy, the AST and ALT >=5 times ULN;
6. For patients with brain metastases, bone metastases or pleural effusion, systemic chemotherapy is proposed after the effective local treatment to control symptoms;
7. Informed consent.

Exclusion criteria:

1. Clinically significant hepatic dysfunction: AST or ALT > 2.5 times the ULN, total serum bilirubin levels > 1.5 times the ULN; clinically significant renal insufficiency: serum creatinine > 1.5 times the ULN;
2. Severe heart disease: New York Heart Association class Ⅲ-IV class of heart failure, unstable angina, myocardial infarction, coronary revascularization six months before randomization;
3. Spleen resection or combined with other severe hematopoietic system diseases;
4. Uncontrolled diabetes, hypertension (above 180/120mmHg), infection or severe gastrointestinal ulcers;
5. History or present with other cancer, except for non melanoma skin cancer, cervical cancer in situ and other cured cancer for at least 5 years;
6. Mental illness, without legal capacity or limited capacity;
7. Pregnancy, lactation or patients with pregnancy plan;
8. Participated in other clinical trail in the past 1 months or participating in other trail now;
9. Other unsuitable condition decided by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520 (Estimated)
Dates: Start 2014-08; Primary Completion 2016-09 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Functional Assessment of Cancer Therapy-Lung scale | 84day
Lung Cancer Symptom Scale | 84day

SECONDARY OUTCOMES:
Anti-cancer drugs common grading evaluation of adverse reaction | 84day
Completion of chemotherapy | 84 day
Objective response rate | 84day
Progression-free survival | 84 day

CONTACTS AND LOCATIONS:
Overall Officials: Jinming Yu, PhD, Study Chair — Shandong Cancer Hospital and Institute; Jie Wang, PhD, Study Chair — Biejing Cancer Hospital